CLINICAL TRIAL: NCT00249821
Title: Optimization of the Dosage Regimen With Growth Hormone Therapy in Children Born Small for Gestational Age. An Open Label, Randomized, Pilot Study, Comparing in Children Treated for 3 Years, the Efficacy of a Saizen® Treatment at the Same Dose Versus a Lower Maintenance Dose Prolonged During 1 Additional Year.
Brief Title: Optimization of the Dosage Regimen of Growth Hormone Therapy in Children Born Small for Gestational Age
Acronym: SGA OPTIMIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono S.A.S., an affiliate of Merck KGaA, Darmstadt, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMP 25735
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Results first posted 2012-10-10 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-08

CONDITIONS: Small Gestational Age (SGA)
MeSH Terms: interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saizen® 0.057 mg/kg/day (Experimental): Subjects who met all inclusion/exclusion criteria were randomly assigned to 0.057 mg/kg/day in this multi-center study. Subjects were stratified at randomization according to the Height-Standard Deviation Score (H-SDS) at this time (less than [<] -2 SDS or greater than [>] -2 SDS)
  Interventions: Drug: Saizen®
- Saizen® 0.035 mg/kg/day (Experimental): Subjects who met all inclusion/exclusion criteria were randomly assigned to 0.035 mg/kg/day in this multi-center study. Subjects were stratified at randomization according to the H-SDS at this time (< -2 SDS or > -2 SDS)
  Interventions: Drug: Saizen®

INTERVENTIONS:
Drug: Saizen® — Saizen® [somatropin (recombinant deoxyribonucleic acid [rDNA] origin) for injection], a r-hGH, is indicated for the treatment of children with growth failure due to inadequate secretion of endogenous growth hormone.
  Other Names: somatropin
  Arms: Saizen® 0.057 mg/kg/day
Drug: Saizen® — Saizen® [somatropin (rDNA origin) for injection], a r-hGH, is indicated for the treatment of children with growth failure due to inadequate secretion of endogenous growth hormone.
  Other Names: somatropin
  Arms: Saizen® 0.035 mg/kg/day

SUMMARY:
Multicentric, open-label, randomized, pilot comparative study in parallel groups comparing 1 group of subjects receiving 0.057 milligram/kilogram/day (mg/kg/day) or 0.40 mg/kg/week of Saizen® during 1 year to 1 group receiving 0.035 mg/kg/day (0.24 mg/kg/week) of Saizen® during 1 year after an initial 3-year treatment of recombinant human growth hormone (r-hGH) therapy with 0.057 mg/kg/day in both groups.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion / randomization into this study, the subjects must fulfill all of the following criteria (if there is no inclusion phase, the inclusion criteria will be considered as inclusion criteria for randomization):

* Written consent form signed by the parents / legal guardian, and child if possible
* Subject born SGA and receiving a r-hGH therapy for this pathology
* Recombinant human growth hormone (r-hGH) started at the maximal chronological age of 7 years for girls and 8 years for boys
* Treatment with r-hGH started for at least 30 months and less than 36 months at 0.057 mg/kg/day
* Height gain during the first 2 years of GH treatment > 1 SD compared with the initial value

Exclusion Criteria:

To be eligible for inclusion in this study the subjects must not meet any of the following criteria:

* Known hypersensitivity to Somatropin or any of the excipients
* Active neoplasia (either newly diagnosed or recurrent)
* Intracranial hypertension
* Known diabetes mellitus
* Proliferative or preproliferative diabetic retinopathy
* Evidence of any progression or recurrence of an underlying intra-cranial space occupying lesion
* Obesity defined as degree 1 on the corpulence curves
* Precocious puberty
* Pubertal status: Tanner breast development stage > 2 for girls, and testicular volume > 4 milliliter (mL) or testicular length > 3 centimeter (cm) and/or testosterone value >1 nanomole/liter [nmol/L] (0.29 gram/mL [g/mL]) for boys For girls > 9 years and Tanner breast development stage 1: uterine size > 35 millimeter (mm)
* Severe chronic concomitant illness such as chronic renal failure, cystic fibrosis
* Concomitant corticoid treatment or levothyroxine treatment other than substitutive treatment, topical or inhaled treatment
* Participation to any clinical study within the 30 days preceding study entry

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2005-02-28 (Actual); Primary Completion 2007-09-30 (Actual); Study Completion 2007-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono S.A.S, France

REFERENCES:
- [Result] Chatelain P, Colle M, Nako JP, Le Luyer B, Wagner K, Berlier P, Tauber M. Optimization of growth hormone dosing in children born small for gestational age: an open-label, randomized study of children during the fourth year of therapy. Horm Res Paediatr. 2012;77(3):156-63. doi: 10.1159/000337216. Epub 2012 Apr 12. PMID 22508151
- See also: Related Info — http://merckserono.com/en/therapeutic_areas/endocrinology/childhood_growth_hormone_defiiency/saizen/saizen.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Saizen® 0.057 mg/kg/Day: Saizen® (recombinant human growth hormone, r-hGH) subcutaneously administered at the daily dose of 0.057 milligram/kilogram (mg/kg) or 0.40 mg/kg/week for duration of 12 months.
- Saizen® 0.035 mg/kg/Day: Saizen® (r-hGH) subcutaneously administered at the daily dose of 0.035 mg/kg or 0.24 mg/kg/week for duration of 12 months.
Period: Overall Study
Arm/Group | Saizen® 0.057 mg/kg/Day | Saizen® 0.035 mg/kg/Day
Started | 10 | 12
Completed | 10 | 11
Not Completed | 0 | 1
Not completed — Technical problem | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saizen® 0.057 mg/kg/Day | Saizen® 0.035 mg/kg/Day | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.00 (1.49) | 7.90 (0.90) | 8.00 (1.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Height Velocity
Description: Height Velocity (HV) is the change in height since the previous year´s measurement and more precisely: HV = {(h-hp)/(d-dp)} * 365.25 [centimeter (cm)/year] where h is current height in cm, hp is previous height in cm, closest to 1 year previous, d is the current date and dp is the date of measurement of previous height, closest to 1 year previous. Additionally, d and dp have to be within 0.6 years and 1.5 years. HV is the mean height velocity over the interval between d and dp but is displayed as HV at d.
Time Frame: Month 12
Population: Full Analysis (FA) set included all the participants who received at least 1 dose of study medication and had at least 1 height evaluation post randomization. Last observation carried forward (LOCF) was used to impute missing values.
Measure: Mean (Standard Deviation); unit: centimeter (cm)/year
Arm/Group | Saizen® 0.057 mg/kg/Day | Saizen® 0.035 mg/kg/Day
Number analyzed (Participants) | 10 | 12
centimeter (cm)/year | 6.40 (1.35) | 4.40 (1.15)
Statistical Analysis 1: Comparison: Saizen® 0.057 mg/kg/Day vs Saizen® 0.035 mg/kg/Day; Month 12: Analysis of co-variance (ANCOVA) method with covariates "height" and "age" at baseline was used to calculate presented p-value; Test type: Superiority or Other; p = 0.001, ANCOVA

2. Secondary Outcome: Change From Baseline in Height-Standard Deviation Score (H-SDS) at Month 6 and Month 12
Description: Height-Standard Deviation Score (H-SDS) was calculated as height minus mean (age-and sex-matched reference) divided by standard deviation (SD) [age and sex-matched reference]. Greater H-SDS indicates greater height.
Time Frame: Baseline (randomization), Month 6 and Month 12
Population: FA set included all the participants who received at least 1 dose of study medication and had at least 1 height evaluation post randomization. LOCF was used to impute missing values.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | Saizen® 0.057 mg/kg/Day | Saizen® 0.035 mg/kg/Day
Number analyzed (Participants) | 10 | 12
standard deviation score
  Baseline (randomization) | -1.30 (0.42) | -1.50 (0.37)
  Change at Month 6 | 0.30 (0.22) | 0.10 (0.10)
  Change at Month 12 | 0.30 (0.30) | -0.10 (0.24)
Statistical Analysis 1: Comparison: Saizen® 0.057 mg/kg/Day vs Saizen® 0.035 mg/kg/Day; Change at Month 6: ANCOVA method with covariates "height" and "age" at baseline was used to calculate presented p-value; Test type: Superiority or Other; p = 0.012, ANCOVA
Statistical Analysis 2: Comparison: Saizen® 0.057 mg/kg/Day vs Saizen® 0.035 mg/kg/Day; Change at Month 12: ANCOVA method with covariates "height" and "age" at baseline was used to calculate presented p-value; Test type: Superiority or Other; p = 0.002, ANCOVA

3. Secondary Outcome: Height Velocity-Standard Deviation Score (HV-SDS)
Description: Height Velocity-Standard Deviation Score (HV-SDS) was calculated as height velocity minus reference mean height velocity divided by SD of the reference mean height velocity. Greater HV-SDS indicates greater height velocity.
Time Frame: Month 6 and Month 12
Population: FA set included all the participants who received at least 1 dose of study medication and had at least 1 height evaluation post randomization. Here "n" signifies number of participants analyzed at that particular time point for each arm group respectively. LOCF was used to impute missing values.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | Saizen® 0.057 mg/kg/Day | Saizen® 0.035 mg/kg/Day
Number analyzed (Participants) | 10 | 12
standard deviation score
  Month 6 (n= 10,11) | 0.60 (0.44) | 0.10 (0.22)
  Month 12 (n=10,12) | 0.30 (0.29) | -0.10 (0.24)
Statistical Analysis 1: Comparison: Saizen® 0.057 mg/kg/Day vs Saizen® 0.035 mg/kg/Day; Month 6: ANCOVA method with covariates "height" and "age" at baseline was used to calculate presented p-value; Test type: Superiority or Other; p = 0.022, ANCOVA
Statistical Analysis 2: Comparison: Saizen® 0.057 mg/kg/Day vs Saizen® 0.035 mg/kg/Day; Month 12: ANCOVA method with covariates "height" and "age" at baseline was used to calculate presented p-value; Test type: Superiority or Other; p = 0.002, ANCOVA

4. Secondary Outcome: Change From Baseline in Height at Month 6
Time Frame: Baseline (randomization) and Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Saizen® 0.057 mg/kg/Day | Saizen® 0.035 mg/kg/Day
Number analyzed (Participants) | 10 | 12
cm
  Baseline (randomization) | 121.10 (7.99) | 119.20 (5.29)
  Change at Month 6 | 3.60 (1.31) | 2.50 (0.99)
Statistical Analysis 1: Comparison: Saizen® 0.057 mg/kg/Day vs Saizen® 0.035 mg/kg/Day; Change at Month 6: ANCOVA method with covariates "height" and "age" at baseline was used to calculate presented p-value; Test type: Superiority or Other; p = 0.029, ANCOVA

5. Secondary Outcome: Change From Baseline in Bone Age at Month 12
Description: Bone age was assessed by a left wrist X-Ray and evaluated by the investigator according to the Greulich and Pyle method.
Time Frame: Baseline (randomization) and Month 12
Population: FA set included all participants who received at least 1 dose of study medication and had at least 1 height evaluation post randomization. 'N' (Number of participants analyzed) signified those participants who were evaluable for this measure and "n" = number of participants analyzed at that particular time point for each arm group respectively.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Saizen® 0.057 mg/kg/Day | Saizen® 0.035 mg/kg/Day
Number analyzed (Participants) | 9 | 10
years
  Baseline (randomization) (n = 9,10) | 7.50 (0.82) | 7.00 (1.85)
  Change at Month 12 (n=9,7) | 1.40 (0.79) | 1.40 (0.89)
Statistical Analysis 1: Comparison: Saizen® 0.057 mg/kg/Day vs Saizen® 0.035 mg/kg/Day; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.972, ANCOVA

6. Secondary Outcome: Insulin Like Growth Factor-1 (IGF-1) Levels
Time Frame: Baseline (randomization), Month 6 and Month 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: microgram/liter (mcg/L)
Arm/Group | Saizen® 0.057 mg/kg/Day | Saizen® 0.035 mg/kg/Day
Number analyzed (Participants) | 10 | 11
microgram/liter (mcg/L)
  Baseline (randomization) (n= 10,11) | 319.60 (146.27) | 275.40 (98.82)
  Month 6 (n= 9,7) | 369.30 (120.13) | 262.40 (65.52)
  Month 12 (n=10,10) | 414.30 (176.70) | 263.00 (120.70)
Statistical Analysis 1: Comparison: Saizen® 0.057 mg/kg/Day vs Saizen® 0.035 mg/kg/Day; Month 6: ANCOVA method with covariates "height" and "age" at baseline was used to calculate presented p-value; Test type: Superiority or Other; p = 0.058, ANCOVA
Statistical Analysis 2: Comparison: Saizen® 0.057 mg/kg/Day vs Saizen® 0.035 mg/kg/Day; Month 12: ANCOVA method with covariates "height" and "age" at baseline was used to calculate presented p-value; Test type: Superiority or Other; p = 0.026, ANCOVA

7. Secondary Outcome: Insulin Like Growth Factor Binding Protein-3 (IGFBP-3) Levels
Time Frame: Baseline (randomization), Month 6 and Month 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: milligram/L (mg/L)
Arm/Group | Saizen® 0.057 mg/kg/Day | Saizen® 0.035 mg/kg/Day
Number analyzed (Participants) | 10 | 10
milligram/L (mg/L)
  Baseline (randomization) (n= 10,10) | 3.40 (0.70) | 3.40 (0.60)
  Month 6 (n= 9,7) | 3.00 (0.84) | 3.30 (0.81)
  Month 12 (n= 9,10) | 3.60 (1.02) | 3.50 (0.77)
Statistical Analysis 1: Comparison: Saizen® 0.057 mg/kg/Day vs Saizen® 0.035 mg/kg/Day; Month 6: ANCOVA method with covariates "height" and "age" at baseline was used to calculate presented p-value; Test type: Superiority or Other; p = 0.793, ANCOVA
Statistical Analysis 2: Comparison: Saizen® 0.057 mg/kg/Day vs Saizen® 0.035 mg/kg/Day; Month 12: ANCOVA method with covariates "height" and "age" at baseline was used to calculate presented p-value; Test type: Superiority or Other; p = 0.055, ANCOVA

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Adverse Events (AEs): Any untoward medical occurrence in the form of signs, clinically significant abnormalities in laboratory findings, diseases, symptoms, or worsening of complications. TEAEs: AEs that occur during treatment with the Investigational Medicinal Product (IMP).
Time Frame: Baseline (randomization) until Month 12
Population: The safety population included all the participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Saizen® 0.057 mg/kg/Day | Saizen® 0.035 mg/kg/Day
Number analyzed (Participants) | 10 | 12
participants | 2 | 1

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected on an ongoing basis from day of written informed consent. All new AEs must be recorded until 4 weeks post drug administration. AEs are classified as pre-treatment, treatment-emergent and post-treatment.
Description: Pre-Treatment:Medical conditions present at initial study visit that did not worsen in severity or frequency during study;Treatment-Emergent: If onset date of AE was on or after the first dose date of the study medication; Post-Treatment: If the onset date of AE was post 4 weeks after drug administration for participants who completed the study.
Arm/Group | Saizen® 0.057 mg/kg/Day | Saizen® 0.035 mg/kg/Day
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 2/10 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saizen® 0.057 mg/kg/Day (N=10) | Saizen® 0.035 mg/kg/Day (N=12)
Asthma (Immune system disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (2) | 0 (0)
Insulin-like growth factor increased (Investigations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Participants' inclusion period was extended but due to remaining low recruitment rate, it was finally decided to stop enrollment even if only 22 participants were enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other